CLINICAL TRIAL: NCT06351293
Title: A Randomized, Split-face Clinical Study on Comparative Analysis of Two Hyaluronic Acid Fillers for Nasolabial Fold Correction
Brief Title: A Comparative Analysis of Two Hyaluronic Acid Fillers for Nasolabial Fold Correction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GLI.04.US.SL.034
Record Dates: First submitted 2024-03-20; First posted 2024-04-08 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2024-10

CONDITIONS: Wrinkle
Keywords: Nasolabial fold

STUDY DESIGN:
Who Masked: Participant
Masking Description: Subjects will be blinded to the treatment assignment, in which randomization and treatment side will be concealed in order to avoid bias in subjective assessment. The clinic staff will mask the product identity by covering the packaging and product name (e.g., using tape, marker, wipe-out, etc.) so that it is not visible to the subjects. The Investigator will not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Defyne Treatment (Experimental): Defyne will be injected into the left or right nasolabial fold, per randomization.
  Interventions: Device: Defyne Treatment in Nasolabial Fold
- RHA3 Treatment (Active Comparator): RHA3 will be injected into the left or right nasolabial fold, per randomization.
  Interventions: Device: RHA3 Treatment in Nasolabial Fold

INTERVENTIONS:
Device: Defyne Treatment in Nasolabial Fold — Defyne will be injected into left or right nasolabial fold, per randomization.
  Arms: Defyne Treatment
Device: RHA3 Treatment in Nasolabial Fold — RHA3 will be injected into left or right nasolabial fold, per randomization.
  Arms: RHA3 Treatment

SUMMARY:
This is a randomized, split-face, subject-blinded, comparative study. Subjects will receive initial treatment with Defyne on one of the NLFs and with RHA3 on the other based on the pre-determined randomization.

4 weeks after the initial treatment, subjects will receive optional touch-up on one side or both sides at the Investigator's discretion for optimal correction.

Subjects to return to the site at Month 3, 6, and 12 for follow-ups.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects 22 to 65 years of age.
2. Subjects with moderate-to-severe NLF based on the 5-point Wrinkle Severity Rating Scale (WSRS), and in the opinion of the investigator, is otherwise a good candidate for treatment with HA fillers.
3. Adult subjects of any gender, race, ethnicity, Fitzpatrick skin type, and sexual orientation.
4. Subjects with general good health.
5. Subjects who are willing to abstain from any other facial plastic surgical or cosmetic procedure(s) during the duration of the study.
6. For female subjects of childbearing potential, she must not be pregnant, breastfeeding or planning pregnancy during the course of the study. Subjects must be willing to take a urine pregnancy test (UPT) prior to all treatments. (Females of non-childbearing potential, e.g., post-menopausal (absence of menstrual bleeding for 1 year without any other medical reason), hysterectomy, or bilateral ovariectomy, are not required to have a UPT.)
7. Subjects who are able and willing to consent to the study informed consent form (ICF), Health Insurance Portability and Accountability Act of 1996 (HIPAA), and photography form prior to any study related procedures.
8. Subjects who agree to be photographed at each visit.
9. Subjects who agree to adhere to the procedures and requirements of the study, to report to the institute on the day(s) and at the time(s) scheduled for the assessments, and to complete all required visits.

Exclusion Criteria:

1. Pregnant, breastfeeding, or planning pregnancy during the course of the study.
2. Current smokers or consumer of nicotine (e.g., cigarettes, e-cigarettes, vaping device with pre-filled pods, vapor tank or mod, chewing tobacco, nicotine replacement therapy).
3. Subjects with history of allergy or hypersensitivity to lidocaine and/or injectable HA.
4. Subjects with previous facial surgery, including aesthetic facial surgical therapy, liposuction, or tattoo in the treatment area.
5. Subjects with previous permanent or semi-permanent implant in proposed treatment area.
6. Subjects with previous biodegradable tissue augmentation therapy in the proposed treatment area within 12 months prior to the baseline visit.
7. Subjects with previous tissue revitalization treatment with neurotoxin in the facial area within 6 months prior to the baseline visit.
8. Subjects with history of other facial treatment/procedure at the study area (NLF) in the previous 6 months that would potentially interfere with study injections (e.g., oral surgery, laser or light therapy, chemical peeling, resurfacing, mesotherapy, dermabrasion).
9. Presence of any disease, lesions, or sign near or on the NLF region, e.g.,

   1. Inflammation, active, or chronic infection in or near the treatment area
   2. Psoriasis, eczema, rosacea, atopic dermatitis, herpes zoster/herpes simplex, and acanthosis
   3. Scars or deformities
   4. Beard or facial hair
10. Subjects with history of bleeding disorders or treatment with anticoagulants or inhibitors of platelet aggregation (e.g., aspirin or other non-steroidal anti-inflammatory drugs), omega 3, or vitamin E within 14 days before treatment. Omega 3 and vitamin E are acceptable only as part of a standard multivitamin formulation.
11. Subjects with tendency to form keloids, hypertrophic scars, or any other healing disorder.
12. Planning on having surgeries and/or invasive medical procedures during the course of the study.
13. Treatment with chemotherapy, immunosuppressive agents, inhaled corticosteroids, immunomodulatory therapy (e.g., monoclonal antibodies or antiviral treatment for human immunodeficiency virus or hepatitis C) within 3 months prior to the baseline visit.
14. Subjects with history of cancer or previous radiation near or on the NLF region.
15. Human immunodeficiency virus positive or active hepatitis.
16. Subjects with any diseases, condition or presentation that may, in the opinion of the investigator, may put the subject at risk, may confound study results, or may interfere with participation in the study.
17. Study site personnel, close relatives of the study site personnel (e.g., parents, children, siblings, or spouse), or employees and close relatives of employees at the Sponsor company.
18. Subjects who have participated in any interventional study within 30 days of enrollment, or subjects planning to participate in any other interventional clinical research study while enrolled in this trial.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2024-02-21 (Actual); Primary Completion 2025-03-17 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Visual Comparison of Nasolabial Fold Ultrasounds | Baseline, Week 4, Month 3, Month 6, Month 12
  A single ultrasound assessment will be taken on each subject's left and right NLF, at neutral expression and at maximum smiling, in photo and video format. The placement of the ultrasound probe will be on the NLF, at the half-way point between nasal ala and oral commissure. Ultrasound assessments will be performed using an 18 MHz GE Venue Fit, a 20 MHz GE, and a 70 MHz Vevo MD ultrasonic transducer interfaced to a system. The probe will have a standard setting of gain, depth, and velocity scale to qualitatively assess placement/depth of filler, size of filler aggregates, and artery in NLF.

SECONDARY OUTCOMES:
Volume Change Imaging Analysis | Baseline, Week 4, Month 3, Month 6, Month 12
  Digital images of the subject's face will be taken of subject's face with a neutral expression and open-mouth maximum smiling expression. These images will be analyzed by VISIA-CRP software for nasolabial fold volume change compared to baseline. A decrease in scores indicates an improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Weiner, MD, Principal Investigator — The Aesthetic Clinique
Locations (1):
- The Aesthetic Clinique, Santa Rosa Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No